CLINICAL TRIAL: NCT02755389
Title: Apneic Oxygenation Via Nasal Cannulae: 15 L/Min vs High-Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Tim Mullen, Staff Anesthesiologist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CapitalDHACanada
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Apneic Oxygenation
Keywords: Tracheal intubation; High flow nasal oxygen; Airway management; Apneic oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0 L/min (Placebo Comparator): These participants will receive 0 L/min oxygen via conventional nasal cannulae during the apneic period.
  Interventions: Drug: 0 L/min oxygen via conventional nasal cannulae
- 15 L/min (Experimental): These participants will receive 15 L/min oxygen via conventional nasal cannulae during the apneic period.
  Interventions: Drug: 15 L/min oxygen via conventional nasal cannulae
- 60 L/min (Experimental): These participants will receive 60 L/min oxygen via high-flow nasal cannulae during the apneic period.
  Interventions: Drug: 60 L/min oxygen via high-flow nasal cannulae

INTERVENTIONS:
Drug: 0 L/min oxygen via conventional nasal cannulae — Patients will have conventional nasal cannulae placed under chin prior to induction of anesthesia. Immediately post-induction these will be placed into the nares. They will be removed from the nares at the end of the study when the airway has been secured. There will be no oxygen flowing through the cannulae in this group during the study.
  Other Names: 0 L/min apneic oxygenation
  Arms: 0 L/min
Drug: 15 L/min oxygen via conventional nasal cannulae — Patients will have conventional nasal cannulae placed under chin prior to induction of anesthesia. Immediately post-induction these will be placed into the nares. They will be removed from the nares at the end of the study when the airway has been secured. There will be 15 L/min of oxygen flowing through the cannulae in this group during the study.
  Other Names: 15 L/min apneic oxygenation
  Arms: 15 L/min
Drug: 60 L/min oxygen via high-flow nasal cannulae — Patients will have high-flow nasal cannulae placed under chin prior to induction of anesthesia. Immediately post-induction these will be placed into the nares. They will be removed from the nares at the end of the study when the airway has been secured. There will be 60 L/min of oxygen flowing through the cannulae in this group during the study.
  Other Names: 60 L/min apneic oxygenation
  Arms: 60 L/min

SUMMARY:
This is a randomized clinical trial investigating the utility of apneic oxygenation via nasal cannulae in the post-induction setting for the purpose of prolonging the safe apneic time. Three groups will be compared, a control group at 0 L/min, a 15 L/min and a 60 L/min group. The primary outcome will be the difference in the partial pressure of oxygen in arterial blood (PaO2) between groups throughout the nine-minute apneic period.

DETAILED DESCRIPTION:
Airway management can be a life saving therapy. One major complication that may occur during airway management is a lack of oxygen in the blood. If severe or prolonged, this lack of oxygen can result in permanent brain damage, damage to other vital organs or even death. Strategies already exist to help prevent a lack of oxygen in the blood (hypoxemia), however research involving new ways to oxygenate patients may help to minimize the chance of hypoxemia during airway management. Apneic oxygenation is a novel method of delivering oxygen to a patient despite a lack of active respiration (i.e. the patient is not breathing on their own and the investigators are not providing the patient an artificial breath). The simplest and least invasive method to provide apneic oxygenation is the application of oxygen through nasal cannulae during airway management. Several different techniques to provide apneic oxygenation via nasal cannulae have been previously described(1-3), however randomized trials comparing these methods do not exist. This study will examine the change over time of the amount of oxygen dissolved in the blood (PaO2) in each of the three treatment groups: a control group (no apneic oxygenation), a 15 L/min group and a 60 L/min group. This data will help to determine the extent of benefit apneic oxygenation provides in this setting.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification 1 to 3
* Body Mass Index 28 to 35
* Elective surgery under general anesthesia

Exclusion Criteria:

* Evidence of difficult airway management (from patient history or clinical examination)
* Features suggestive of difficult bag mask ventilation
* Significant uncontrolled gastroesophageal reflux disease
* Significant respiratory disease (including severe asthma or chronic obstructive pulmonary disease, oxygen dependency, pulmonary hypertension, identified by pulmonary function tests or inability to climb one flight of stairs)
* Significant cardiac disease (ischemic heart disease, severe valvular disease, severe arrhythmia, congestive heart failure, ejection fraction < 50%, inability to climb one flight of stairs)
* Inability to lie flat (skeletal deformities, orthopnea)
* Hemoglobin < 100 g/L
* Pregnancy
* Neuromuscular disorder
* Known or suspected cervical spine instability
* Patients undergoing neurosurgical procedures
* Any clinical or radiological evidence of increased intracranial pressure
* Any expected requirement for rapid sequence intubation
* Allergy to any of the agents used for induction of general anesthesia in the study
* Contraindication to insertion of radial artery cannula
* Uncorrected coagulopathy
* Significant nasal obstruction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
PaO2: repeated measures every 90 seconds after induction | 0-9 minutes after induction
  data collected from serial arterial blood gas measurements

SECONDARY OUTCOMES:
Partial pressure of carbon dioxide in arterial blood (PaCO2): repeated measures every 90 seconds after induction | 0-9 minutes after induction
  data collected from serial arterial blood gas measurements
Lowest oxygen saturation by pulse oximetry (SpO2) encountered during study | 0-9 minutes after induction
  continuous monitoring: data collected from electronic charting software
Time to desaturation below 95% SpO2 | 0-9 minutes after induction
  continuous monitoring: data collected from electronic charting software
Number of participants with SpO2 below 95% | 0-9 minutes after induction
  continuous monitoring: data collected from electronic charting software

OTHER OUTCOMES:
Number of participants with sore throat | 1 hour post-operative or transfer out of post-anaesthesia care unit (PACU) if less than 1 hour post-operative
  Data collected with PACU nurse questionnaire
Number of participants with nausea | 1 hour post-operative or transfer out of PACU if less than 1 hour post-operative
  Data collected with PACU nurse questionnaire
Number of participants with epistaxis | 1 hour post-operative or transfer out of PACU if less than 1 hour post-operative
  Data collected with PACU nurse and staff anesthesiologist questionnaires
Number of participants with gastroesophageal regurgitation prior to endotracheal tube (ETT) placement | Assessed at 90 seconds and 9 minutes after induction
  Data collected with staff anesthesiologist questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mullen, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Halifax Infirmary, QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000
- [Background] Christodoulou C, Rohald P, Mullen T. (2013). Apneic oxygenation via nasal prongs at 10 L/min prevents hypoxemia during tracheal intubation for elective surgery. European Respiratory Society Annual Congress 2013. Abstract Number: 5356 Publication Number: P4923